CLINICAL TRIAL: NCT00067782
Title: A Phase IIIB Study Evaluating the Effect on Serum Lipids Following a Switch to Atazanavir in HIV Infected Subjects Evidencing Virologic Suppression on Their First PI-Based Antiretroviral Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AI424-067
Record Dates: First submitted 2003-08-27; First posted 2003-08-28 (Estimated); Last update posted 2011-04-14 (Estimated); Status verified 2010-01

CONDITIONS: HIV Infections
Keywords: HIV; Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — Atazanavir Sulfate

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Atazanavir (immediate switch)
- 2 (Active Comparator)
  Interventions: Drug: Atazanavir (Week 24 switch)

INTERVENTIONS:
Drug: Atazanavir (immediate switch) — Capsules, Oral, 400mg, Once daily, 48 weeks.
  Other Names: Reyataz
  Arms: 1
Drug: Atazanavir (Week 24 switch) — Capsules, Oral, 400mg, Once daily, 48 weeks.
  Other Names: Reyataz
  Arms: 2

SUMMARY:
The purpose of this clinical research study is to learn if atazanavir is associated with serum LDL cholesterol in HIV-infected subjects following a substitution of atazanavir for their previously administered protease inhibitor.

ELIGIBILITY:
Key Inclusion Criteria:

* Must be on current HIV treatment regimen at least 3 to 6 months prior to study (this must be one protease inhibitor, or ritonavir-boosted protease inhibitor, and two nucleoside reverse transcriptase inhibitors) must be subject's first PI ever received
* Plasma HIV-1 RNA level < 50 c/mL within 3 to 6 months prior to study start
* Fasting LDL cholesterol > 130 mg/dL

Key Exclusion Criteria:

* WOCBP who do not use effective barrier contraception for any reason
* Women who are pregnant or breast feeding
* A life expectancy < 12 months
* Presence of a newly diagnosed HIV-related OI or any medical condition requiring acute therapy at the time of enrollment
* Cushing's Syndrome
* Uncontrolled diabetes mellitus, history of diabetic ketoacidosis or hyperosmolar syndrome
* Untreated hypothyroidism or hyperthyroidism
* Nephrotic syndrome or significant proteinuria
* Obstructive liver disease
* Active alcohol or substance abuse
* Proven or suspected acute hepatitis in the 30 days prior to study entry
* Intractable diarrhea (greater than or equal to 6 loose stools/day for at least 7 consecutive days) within 30 days prior to study start
* History of acute or chronic pancreatitis
* Inability to swallow capsules
* Presence of cardiomyopathy
* Known history of prolonged QTc interval
* Any of the following:

  1. clinical symptoms potentially related to heart block
  2. heart rate < 40 bpm
  3. any of the following EKG abnormalities:

  i) pause length > 3 seconds ii) second or third degree AV heart block iii) QTc interval > 450 msec for males iv) QTc interval > 470 msec for females
* Fasting serum triglyceride level > 750 mg/dL
* Any of the following lab values within 2 weeks of starting study drug:

  1. serum creatinine greater to or equal to 1.5 times the upper limit of normal
  2. total serum lipase greater than or equal to 1.4 times the upper limit of normal
  3. liver transaminases greater than or equal to 3 times the upper limit of normal
  4. total serum bilirubin greater than or equal to 1.5 times the upper limit of normal
* Hypersensitivity to any component of the formulation of study drug
* Use of any lipid-lowering agent within 4 weeks prior or during study
* Use of a PI-containing ARV regimen prior to entry which is comprised of more than one PI
* Inclusion of an NNRTI in the PI-containing regimen
* Prisoners or subjects involuntary incarcerated for treatment of psychiatric or physical illness

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2002-12; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Time to virologic rebound for subjects with HIV RNA < 50 c/mL at baseline; Magnitude/ durability of increases from baseline in absolute CD4 (Time-Averaged Difference) through WK12; Mean % change from baseline in fasting LDL cholesterol at WK12.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (19):
- United States (19):
  - Local Institution, Phoenix, Arizona
  - Local Institution, West Hollywood, California
  - Local Institution, Washington D.C., District of Columbia
  - Local Institution, Altamonte Springs, Florida
  - Local Institution, Fort Lauderdale, Florida
  - Local Institution, Miami, Florida
  - Local Institution, Tampa, Florida
  - Local Institution, Boston, Massachusetts
  - Local Institution, Minneapolis, Minnesota
  - Local Institution, St Louis, Missouri
  - Local Institution, East Orange, New Jersey
  - Local Institution, New York, New York
  - Local Institution, Huntersville, North Carolina
  - Local Institution, Cleveland, Ohio
  - Local Institution, Oklahoma City, Oklahoma
  - Local Institution, Philadelphia, Pennsylvania
  - Local Institution, Columbia, South Carolina
  - Local Institution, Fort Worth, Texas
  - Local Institution, Houston, Texas